CLINICAL TRIAL: NCT01321905
Title: 5-month Pilot Intervention Study on Vitamin D in Patients With Cystic Fibrosis
Brief Title: Prospective Intervention Study on Vitamin D in Patients With Cystic Fibrosis
Acronym: D-vitamin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Terezia Pincikova, Pulmonologist, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/1723-31/1
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ergocalciferol (Experimental): Patients younger than 16 years of age are administered 35,000 IU ergocalciferol per week divided into doses 5000 IU per day as a starting dose that is further adjusted by serum 25-hydroxy vitamin D concentration monitoring.
  Patients 16 or more years of age are administered 50,000 IU ergocalciferol per week divided into doses 7150 IU per day as a starting dose that is further adjusted by serum 25-hydroxy vitamin D concentration monitoring.
  Interventions: Dietary Supplement: Supplementation with vitamin D2/D3
- Cholecalciferol (Experimental): Patients younger than 16 years of age are administered 35,000 IU cholecalciferol per week divided into doses 5000 IU per day as a starting dose that is further adjusted by serum 25-hydroxy vitamin D concentration monitoring.
  Patients 16 or more years of age are administered 50,000 IU cholecalciferol per week divided into doses 7150 IU per day as a starting dose that is further adjusted by serum 25-hydroxy vitamin D concentration monitoring.
  Interventions: Dietary Supplement: Supplementation with vitamin D2/D3
- Control (No Intervention): Patients continue their ordinary vitamin supplementation without getting extra vitamin D supplements.

INTERVENTIONS:
Dietary Supplement: Supplementation with vitamin D2/D3 — Patients younger than 16 years of age are administered 35,000 IU ergo-/chole-calciferol per week divided into doses 5000 IU per day as a starting dose that is further adjusted by serum 25-hydroxy vitamin D concentration monitoring. The intervention time is 3 months, followed by 2-months wash-out period when patients do not take any more extra vitamin D but they are still monitored.
  Patients 16 or more years of age are administered 50,000 IU ergo-/chole-calciferol per week divided into doses 7150 IU per day as a starting dose that is further adjusted by serum 25-hydroxy vitamin D concentration monitoring.
  Arms: Cholecalciferol; Ergocalciferol

SUMMARY:
The vast majority of Cystic Fibrosis (CF) patients worldwide are vitamin D insufficient. There is no evidence of benefit of vitamin D supplementation for CF patients yet. However, descriptive cross-sectional studies suggest that vitamin D might be beneficial with respect to bone health, as well as to the newly described "non-classical" functions of vitamin D such as the potential anti-diabetic and immunomodulatory effects. To prove causation, and to determine which serum vitamin D concentration is optimal for CF patients, vitamin D supplementation interventional studies are needed, such as our trial.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of cystic fibrosis
* Age 6 years and more
* Serum 25-hydroxy vitamin D concentration at the latest visit < 75 nmol/L

Exclusion Criteria:

* Pregnancy or lactation
* Established diagnosis of CF-related diabetes
* CF-related liver disease
* Status post transplantation (lung, liver or other)
* Long-term corticosteroid treatment per os
* Hypercalcaemia or kidney stones
* Use of tanning beds more often than once a month
* At inclusion, plans to travel to a sunny location for more than 1 week during the study period
* Any known disorders of the endocrine system affecting vitamin D metabolism (hyperparathyroidism, malignancy, advanced renal disease)
* Inclusion into another study testing immunomodulatory substances

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Serum 25-hydroxy vitamin D | 3 months
  This pilot study is primarily designed for establishing effective vitamin D dosing in our specific patient population, and only secondarily designed (and thus, not powered for) for the secondary outcome measures. The results of this study will make it possible for the first time to power the follow-up long-term study for some of the secondary outcome measures followed in this pilot study, some of which might therefore become primary outcome measures in the follow-up study.

SECONDARY OUTCOMES:
Parathyroid hormone (PTH) | 3 months
  As a surrogate marker of bone health
Inflammatory parameters | 3 months
  Cytokine profiles, antimicrobial peptides, peripheral blood mononuclear cell profiles, immunoglobulines, acute phase markers, sedimentation rate and other
Infection parameters | 3 months
  Number of days on intravenous antibiotic treatment; number of infectious episodes; number of common cold episodes; relative number of sputum samples positive for pathological bacteria; and other
Lung function parameters | 3 months
  FEV1, FVC, PEF, FEF25, FEF50, FEF75 and other
Glucose tolerance parameters | 3 months
  Insulin, C-peptide, glucagon, fasting plasma glucose, HbA1c, 3-hour 75-g oral glucose tolerance test
Adherence with vitamin D treatment | 3 months
  Semi-quantitative assessment by a questionnaire (thus, a patient-reported outcome)
Disease-specific quality of life | 3 months
  Assessment using "CFQ-R" questionnaire, specifically designed to measure the quality of life in CF patients
Plasma calcium | 3 months
  Proportion of patients with albumin-corrected serum calcium increasing to a concentration greater than 2,75 mmol/L in patients with no hypercalcaemia before vitamin D supplementation was started.
Relative number of patients reaching high abnormal 25(OH)D concentrations | 3 months
  Proportion of patients in the intervention arms reaching 25(OH)D >250 nmol/L
Proportion of patients reaching toxic 25(OH)D concentrations | 3 months
  Proportion of patients in the intervention arms reaching 25(OH)D >375 nmol/L
Proportion of patients with suspect hypercalcaemia symptoms | 3 months
  Proportion of patients with suspect hypercalcaemia symptoms in the intervention arms

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm Cystic Fibrosis Center, Karolinska University Hospital Huddinge, Stockholm, Sweden

REFERENCES:
- [Derived] Pincikova T, Paquin-Proulx D, Sandberg JK, Flodstrom-Tullberg M, Hjelte L. Vitamin D treatment modulates immune activation in cystic fibrosis. Clin Exp Immunol. 2017 Sep;189(3):359-371. doi: 10.1111/cei.12984. Epub 2017 May 24. PMID 28470739
- [Derived] Pincikova T, Paquin-Proulx D, Sandberg JK, Flodstrom-Tullberg M, Hjelte L. Clinical impact of vitamin D treatment in cystic fibrosis: a pilot randomized, controlled trial. Eur J Clin Nutr. 2017 Feb;71(2):203-205. doi: 10.1038/ejcn.2016.259. Epub 2016 Dec 14. PMID 27966575